CLINICAL TRIAL: NCT05565755
Title: Impact on Patients' Vaccine Hesitancy of a Motivational Interviewing Training in Initial Medical Training Course
Acronym: MOTI-VAC_IMG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2020-15
Record Dates: First submitted 2022-09-26; First posted 2022-10-04 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: Vaccination Hesitancy
MeSH Terms: conditions — Vaccination Hesitancy | interventions — Motivational Interviewing

STUDY DESIGN:
Intervention Model Description: Comparison of vaccine hesitancy in parents of adolescents during consultations by 2 different groups of interns:
  * a group of interns trained in MI
  * a group of interns not trained in IM The randomization will be done by random draw from the 3rd year list of general medicine interns.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Parents of adolescents who had a consultation with a group of IM-trained interns. (Experimental)
  Interventions: Other: Motivational interview
- Parents of adolescents who have not had a consultation with a group of IM trained interns. (No Intervention)

INTERVENTIONS:
Other: Motivational interview — Motivational interview Training
  Arms: Parents of adolescents who had a consultation with a group of IM-trained interns.

SUMMARY:
In France, vaccination coverage of adolescents remains suboptimal, partly because of a loss of confidence, favoring the re-emergence of epidemics. Despite the extension of mandatory vaccination, some vaccines are still recommended.

Motivational Interviewing (MI), which reinforces a person's own motivation and commitment to change, has been shown to be effective in addiction, nutrition, physical activity and vaccination (Promovac study in Quebec). However, it has not been evaluated in the French cultural context (with mandatory vaccination).

The main objective will be to measure the effect of training in MI for general medical interns at the end of their studies on the vaccine hesitancy (VH) of parents of adolescents consulting in primary care, using a validated scale: VCS.

A multicenter study will be conducted in two university departments of general medicine (Marseille and Nice), comparative, clustered exposure/non-exposure type. It will compare the HV of parents of adolescents during consultations by 2 different groups of interns:

* a group of interns trained in MI,
* a group of interns not trained in MI. The randomization will be done by random draw from the 3rd year list of GP interns not in SASPAS training.

After the MI training, each intern in the "exposed" and "unexposed" groups will have 4 months to include at least 3 parents of adolescents seen in consultation.

Descriptive analyses will be performed followed by statistical analysis by modeling the standardized HV score using hierarchical linear regression.

Training of interns in MI applied to vaccination will increase their knowledge, skills and confidence in using this technique.

We can expect a decrease in VH among parents in primary care who consulted a physician trained in MI.

ELIGIBILITY:
Inclusion Criteria:

* Interns who are not in SASPAS for the semester from early November 2020 to the end of April 2021 and who will complete the SASPAS internship in the following semester (May 2021 to October 2021).

Exclusion Criteria:

* Intern on availability or inter-CHU internship for the semester November 2020 to end of April 2021
* Interns who have already received training at the MI

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2020-07-15 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-08-08 (Estimated)

PRIMARY OUTCOMES:
Vaccine hesitancy score of parents of adolescents | through study completion, an average of 2 years
  Score measured using the validated VCS: Vaccination Confidence Scale. This scale is composed of 8 items, each receiving a score ranging from 0 (strongly disagree) to 10 (strongly agree), with the highest score expressing the highest degree of confidence in vaccines and the lowest expressing the highest degree of VH.

SECONDARY OUTCOMES:
Behaviour, beliefs and knowledge about vaccines | through study completion, an average of 2 years
  Reponses to Questions about Behaviour, beliefs and knowledge about vaccine
Parent and medical intern satisfaction with the consultation | through study completion, an average of 2 years
  Level of parent satisfaction on a scale (not very satisfied to very satisfied)
MI learning, knowledge and skills for vaccination promotion in interns | year 2
  Score to the motivational interviewing skills in immunization Questionnaire (MISI)

CONTACTS AND LOCATIONS:
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: Undecided